CLINICAL TRIAL: NCT07297433
Title: Erector Spinae Plane Block in Laparoscopic Colorectal Cancer Surgery: Effects on Renal Blood Flow and Kidney Function
Brief Title: Erector Spinae Plane Block in Laparoscopic Colorectal Cancer Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, Arif Enes Koyuncu, Research assistant doktor, Kayseri City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KayseriCH-AAR-AEK-01
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Kolon Kanseri
Keywords: Erector spinae plane block; Laparoscopic surgery; Near-infrared spectroscopy; Postoperative kidney injury; Colorectal cancers
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be randomized using the sealed envelope method. The anesthesiologist performing the procedure will be fixed, and the person keeping records will always be another anesthesiologist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients will be informed about the operation and the procedure to be performed during a preoperative consultation. Patients included in the study will be taken to the operating room after reading and signing the informed consent form. Bilateral erector spinae plane block will be administered to patients in this group prior to surgery. Renal blood flow will be monitored using NIRS. Postoperative period: NGAL, serum creatinine, and eGFR values will be measured at 2, 6, and 24 hours.
  Interventions: Other: Erector Spinae Plane Block
- Control group (No Intervention): Patients will be interviewed before surgery and informed about the surgery and the procedure to be performed. Patients to be included in the study will be taken to the operating room after reading and approving the informed consent form. Patients in this group will not undergo erector spinae plane block. Renal blood flow will be monitored using NIRS. In the postoperative period, NGAL, serum creatinine, and eGFR values will be measured at 2, 6, and 24 hours.

INTERVENTIONS:
Other: Erector Spinae Plane Block — The erector spinae plane block (ESP) is a block that is easy to perform with ultrasound (USG) guidance and has a relatively low risk of mechanical complications. It has quickly become popular and is used in various indications in anesthesiology and resuscitation clinics.
  Arms: Intervention group

SUMMARY:
Our study will compare patients who underwent laparoscopic surgery for colorectal cancer with and without Erector Spinae Plane Block in terms of renal blood flow and renal function tests. In our study, which will be conducted by dividing patients into two groups, the investigators aim to demonstrate the effects of the erector spinae plane block on renal physiology by simultaneously monitoring renal blood flow during the intraoperative period using near-infrared spectroscopy and monitoring renal function in the postoperative period using NGAL, serum creatinine, and eGFR.

DETAILED DESCRIPTION:
Our study comparing patients who did and did not undergo ESBP in terms of renal blood flow and renal function tests during laparoscopic surgeries for colorectal cancer is planned to be conducted at Kayseri City Hospital with volunteer patients.

The erector spinae plane block (ESP) is a block that is easy to perform with ultrasound (USG) guidance and has a relatively low risk of mechanical complications. It has quickly become popular and is used in various indications in anesthesiology and resuscitation clinics.

The total number of volunteers expected to participate in this study is 60. Patients will be randomly assigned to two groups using a sealed envelope method. The number of volunteers determined for each group is 30.

Patients will be interviewed before the operation and informed about the operation and the procedure to be performed. After reading and approving the informed consent form, patients to be included in the study will be divided into two groups using the sealed envelope method. Group 1 will receive ESP block, while Group 2 will be the control group and will not receive any block.

All patients will be monitored throughout the operation using invasive blood pressure, ECG, and pulse oximetry. Following preoxygenation, induction will be administered with intravenous propofol (2 mg/kg), fentanyl 1 µg/kg, and rocuronium (0.6 mg/kg) injections. After tracheal intubation, an arterial catheter will be placed in the radial artery to continuously monitor blood pressure. Anesthesia maintenance will be achieved with inhaled sevoflurane and intravenous remifentanil infusion. After induction, patients will be placed in the left-right lateral decubitus position, and bilateral blocks will be performed with ultrasound guidance.

Group 1: ESP block, 0.5% bupivacaine 0.2-0.4 ml/kg will be administered. Group 2: Patient group without block.

After ESBP application, the 'Near infrared spectroscopy' device will be placed on the bilateral 9-10th posterior costal region (flank region) of the patients in a manner suitable for observing renal blood flow. Monitoring will be performed throughout the operation and recorded on the follow-up form. N-GAL, serum creatinine, and eGFR values will be measured in both groups during the preoperative and postoperative periods (at 2, 6, and 24 hours).

Once the expected number of patients is reached, the data obtained will be statistically evaluated and recorded.

After the data is collected, it will be processed for statistical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age: 35-75 years old
* Colorectal cancer surgery must be planned by a physician
* No infection in the injection site
* No history of any disease related to clotting or bleeding time
* The patient must be a volunteer
* No history of local anesthetic allergy

Exclusion Criteria:

* Being under 18 years of age
* Having a systemic infection or infection at the injection site
* Having any disease related to bleeding time and clotting
* Having a history of local anesthetic allergy
* Patient refusal (ESPB for analgesic purposes)
* Patients with a Body Mass Index (BMI) of 30 or above

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-05 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Neutrophil gelatinase-associated lipocalin (NGAL) | For 24 hours after procedure
  Neutrophil gelatinase-associated lipocalin (NGAL) is a small, stable protein synthesized by various epithelia, including neutrophils and renal proximal tubules. Its dramatic increase in urine following kidney injury has made NGAL a useful biomarker for kidney damage today. According to the catalog information, serum NGAL kits can measure between 15-1300 ng/ml. Values above 150 ng/ml are considered positive. Results above 170 ng/ml in adult patients and above 100-135 ng/ml in pediatric patients are considered positive.
Serum Kreatinin | For 24 hours after the procedure
  In adults, the normal range for creatinine is generally 0.7 to 1.2 milligrams per deciliter (mg/dL) for men and 0.5 to 0.9 mg/dL for women. Reference ranges may vary between laboratories.
eGFR | For 24 hours after the procedure
  EGFR>90: Minimal kidney damage based on normal GFR or urine test results EGFR between 60-89: Mild decrease in GFR EGFR between 30-59: Moderate decrease in GFR EGFR between 15-29: Severe decrease in GFR EGFR<15: Kidney failure
Near-Infrared Spectroscopy (NIRS) | During the operation period
  Near-Infrared Spectroscopy (NIRS) is a non-invasive method for assessing tissue oxygenation. It is increasingly used to monitor renal perfusion, particularly in critically ill patients, during surgery, and in intensive care units, where it is important for evaluating kidney oxygenation. NIRS measures the absorption of near-infrared light (700-1000 nm) sent to the tissue by the oxygenated (HbO₂) and deoxygenated (Hb) forms of hemoglobin. In laparoscopic surgeries, renal blood flow may decrease without a drop in blood pressure, and acute kidney injury may occur in the postoperative period. NIRS is used to predict this condition.

CONTACTS AND LOCATIONS:
Overall Officials: Günhan Gökahmetoğlu, Principal Investigator — Kayseri City Hospital
Locations (1):
- Kayseri Şehir Hastanesi, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No